CLINICAL TRIAL: NCT02137343
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled Study of Rilotumumab (AMG 102) With Cisplatin and Capecitabine (CX) as First-line Therapy in Advanced MET-Positive Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Phase 3 Study of Rilotumumab (AMG 102) With Cisplatin and Capecitabine (CX) as First-line Therapy in Gastric Cancer
Acronym: RILOMET-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: All Amgen sponsored AMG102 clinical studies were terminated following a pre-planned Data Monitoring Committee safety review of study 20070622.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120142
Record Dates: First submitted 2014-04-28; First posted 2014-05-13 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; First Line Treatment Gastroesophageal Junction (GEJ); Gastroesophageal Junction Cancer (GEJ); GEJ Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — rilotumumab; Cisplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilotumumab (Experimental): Rilotumumab plus Cisplatin and Capecitabine (CX).
  Interventions: Drug: Rilotumumab; Drug: Cisplatin; Drug: Capecitabine
- Placebo (Placebo Comparator): Rilotumumab-placebo plus Cisplatin and Capecitabine (CX).
  Interventions: Drug: Placebo; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Rilotumumab — Rilotumumab is a fully human monoclonal antibody immunoglobulin G, type 2 (IgG2) against human hepatocyte growth factor/scatter factor (HGF/SF) that blocks binding of HGF/SF to its receptor MET, inhibiting HGF/SF/MET-driven activities in cells.
  Other Names: AMG102
  Arms: Rilotumumab
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Cisplatin — A platinum containing chemo-therapy compound that reacts in vivo, binding to and causing crosslinking of DNA, which ultimately triggers apoptosis (programmed cell death)
  Other Names: Platinol; Platinal-AQ
Drug: Capecitabine — A chemo-therapy prodrug that is enzymatically converted to 5-fluorouracil in the tumor, where it inhibits DNA synthesis and slows growth of tumor tissue.
  Other Names: Xeloda

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo controlled study of Rilotumumab (AMG 102) with Cisplatin and Capecitabine (CX) for untreated advanced mesenchymal epithelial transition factor (MET)-positive gastric or gastroesophageal junction adenocarcinoma (GEJ).

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically confirmed unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Tumor MET-positive by immunohistochemistry (IHC).
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Male or female subject greater than or equal to 20 years of age at the time of informed consent.

Key Exclusion Criteria:

* Human epidermal growth factor receptor 2 (HER2)-overexpressing locally advanced or metastatic gastric or GEJ adenocarcinoma.
* Previous systemic therapy for locally advanced or metastatic gastric or GEJ or lower esophageal adenocarcinoma.
* Less than 6 months have elapsed from completion of prior neoadjuvant or adjuvant chemotherapy or chemoradiotherapy to randomization.
* Squamous cell histology.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 4 years
  To determine if the treatment of rilotumumab in combination with CX significantly improves progression-free survival as compared with rilotumumab-placebo in combination with CX in subjects with unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma with MET-positive expression.
Overall Survival | 4 years
  To determine if the treatment of rilotumumab in combination with CX significantly improves overall survival as compared with rilotumumab-placebo in combination with CX in subjects with unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma with MET-positive expression.

SECONDARY OUTCOMES:
TTP | 4 years
  Time to Progression (TTP)
ORR | 4 years
  Objective Response Rate
DCR | 4 years
  Disease Control Rate
TTR | 4 years
  Time to Response
Incidence of subject adverse events, laboratory abnormalities and immunogenicity | 4 years
  Adverse events and laboratory abnormalities are reported by Common Terminology Criteria for Adverse Events (CTCAE) (v3.0)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- Japan (16):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Kashiwa-shi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi-shi, Hyōgo
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Osaka, Osaka
  - Research Site, Osakasayama-shi, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Takatsuki-shi, Osaka
  - Research Site, Kitaadachi-gun, Saitama
  - Research Site, Suntou-gun, Shizuoka
  - Research Site, Utsunomiya, Tochigi
  - Research Site, Bunkyo-ku, Tokyo
- South Korea (3):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Hwasun
  - Research Site, Seoul

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com